CLINICAL TRIAL: NCT03755102
Title: A Pilot Study of Dacomitinib With or Without Osimertinib for Patients With Metastatic EGFR Mutant Lung Cancers With Disease Progressionon Osimertinib.
Brief Title: A Pilot Study of Dacomitinib With or Without Osimertinib for Patients With Metastatic EGFR Mutant Lung Cancers With Disease Progression on Osimertinib.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-341
Record Dates: First submitted 2018-11-26; First posted 2018-11-27 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2022-11

CONDITIONS: EGFR Gene Mutation; Lung Cancer; Lung Cancer Metastatic
Keywords: EGFR C797S; EGFR mutant lung cancer; dacomitinib; osimertinib; 18-341; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Lung Neoplasms | interventions — dacomitinib; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Participants treated with dacomitinib alone (Experimental): Participants in this cohort have a somatic activating mutation in EGFR in a tumor biopsy or plasma cfDNA liquid biopsy.
  Interventions: Drug: Dacomitinib
- Cohort 2: Participants treated with dacomitinib in combination with osimertinib (Experimental): Participants in this cohort have a secondary acquired EGFR mutation in addition to the sensitizing mutation
  Interventions: Drug: Dacomitinib; Drug: Osimertinib

INTERVENTIONS:
Drug: Dacomitinib — Cohort 1 Dacomitinib Dosing:
  Dose level 1: Dacomitinib 45mg daily Dose level -1: Dacomitinib 30mg daily Dose level -2: Dacomitinib 15mg daily
  Cohort 2 Dacomitinib Dosing:
  Dose level 1: Dacomitinib 30 mg daily Dose level -1: Dacomitinib 15 mg daily
Drug: Osimertinib — In cohort 2, participants will begin on dacomitinib orally daily in combination with Osimertinib
  Dose level Osimertinib Dosing:
  Dose level 1: Osimertinib 80 mg daily Dose level -1: Osimertinib 40 mg daily
  Arms: Cohort 2: Participants treated with dacomitinib in combination with osimertinib

SUMMARY:
The purpose of this study is to assess whether dacomitinib after osimertinib is effective in participants with metastatic EGR-mutant lung cancers.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Advanced biopsy-proven metastatic non-small cell lung cancer
* Somatic activating mutation in EGFR in a tumor biopsy or plasma cfDNA liquid biopsy
* Prior treatment with osimertinib with response followed by disease progression
* No prior first or second generation EGFR inhibitor treatment (gefitinib, afatinib, erlotinib)
* Archival tissue available from a tumor biopsy done after disease progression on osimertinib or willing to undergo a tumor biopsy or liquid biopsy after disease progression on osimertinib prior to study initiation
* Measurable (RECIST 1.1) indicator lesion not previously irradiated
* Karnofsky performance status (KPS) >/= 70%
* Age >/= 18 years old
* Ability to swallow oral medication
* Adequate organ function

  * AST, ALT </= 3 x ULN
  * Total bilirubin </= 1.5x ULN
  * Creatinine </= 1.5x ULN OR calculated creatinine clearance >/= 60ml/min
  * Absolute neutrophil count (ANC) >/= 1000 cells/mm3
  * Hemoglobin>/=8.0 g/dL
  * Platelets >/=75,000/mm3

Exclusion Criteria:

* Pregnant or lactating women
* Any radiotherapy within 1 week of starting treatment on protocol.
* Any major surgery within 1 weeks of starting treatment on protocol.
* Any evidence of active clinically significant interstitial lung disease
* Continue to have unresolved > grade 1 toxicity from any previous treatment Treatment
* Patients with a known mechanism of resistance to osimertinib that will clearly not respond to dacomitinib therapy (i.e. known MET amplification, ALK fusion, RET fusion).
* Symptomatic brain metastases or leptomeningeal disease requiring escalating doses of steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | 1 year
  Overall response rate (partial and complete responses) of dacomitinib in participants with EGFR-mutant lung cancers and disease progression on osimertinib

SECONDARY OUTCOMES:
Progression-free survival | 1 year
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Helen Yu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org